CLINICAL TRIAL: NCT06512402
Title: Epinephrine Versus Norepinephrine Infusion for Prevention of Maternal Hypotension During Caesarean Delivery: a Randomized Clinical Trial
Brief Title: Epinephrine Vs Norepinephrine Infusion During Caesarean Delivery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS-376-2023
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Hypotension; Spinal Block; Cesarean Section
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norepinephrine group (Active Comparator): After subarachnoid block, mothers will be placed in supine position with left-lateral tilt and will receive norepinephrine infusion until 5 min after delivery
  Interventions: Drug: Norepinephrine
- Epinephrine group (Active Comparator): After subarachnoid block, mothers will be placed in supine position with left-lateral tilt and will receive epinephrine infusion until 5 min after delivery
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: Norepinephrine — patients will receive norepinephrine infusion at rate of 0.05 mcg/Kg/min
  Arms: Norepinephrine group
Drug: Epinephrine — patients will receive epinephrine infusion dose of 0.03 mcg/Kg/min
  Arms: Epinephrine group

SUMMARY:
Epinephrine is a well-known vasoactive agent in medical practice. However, its use is obstetric population is still scanty. Few studies evaluated the use of epinephrine during Cesarean delivery and a recent randomized controlled dose-finding trial reached an acceptable incidence of hypotension (13%) with the use of 0.03 mcg/kg/min as prophylaxis.

Being a newly introduced vasoactive agent in obstetric practice, it is essential to be adequately compared with other vasopressors using the optimum dosage and appropriate outcomes.

There are no data, till date, comparing epinephrine versus norepinephrine infusion during Cesarean delivery using a composite outcome of hypotension, hypertension, and bradycardia. The aim of this study is to compare epinephrine versus norepinephrine infusion for prophylaxis against post-spinal hypotension during Caesarean delivery

DETAILED DESCRIPTION:
Upon arrival to the operating room, routine monitoring will be applied (electrocardiography, pulse oximetry, and non-invasive blood pressure monitor). An 18G-cannula will be inserted, and 10 mg metoclopramide, and 50 mg ranitidine will be delivered. Co-load infusion of lactated Ringer's solution will be infused at rate of 15 mL/Kg over 10 minutes; and 10 mg hyperbaric bupivacaine in addition to 20 mcg fentanyl will be injected in the subarachnoid space at L3-L4 or L4-L5 interspace using 25G spinal needle.

After subarachnoid block, mothers will be placed in supine position with left-lateral tilt and will receive the vasopressor infusion according to the allocated study group Block success will be assessed after 5 minutes from injecting local anesthetic into the subarachnoid space using pinprick; and will be confirmed if sensory block level is at T4. The vasopressor will be infused in the same line with intravenous fluids using a three-way stopcock. The baseline systolic blood pressure reading will be calculated as the average of 3 readings obtained in the supine position with left-uterine displacement at two-minute intervals with a difference of <10%.

Hemodynamic management in both groups will be as follow:

Post-spinal hypotension (defined as systolic blood pressure ≤80% of the baseline reading or systolic blood pressure <90 mmHg during the period from intrathecal injection to delivery of the fetus) will be managed by ephedrine 9 mg Severe post-spinal hypotension (defined as systolic blood pressure ≤60% of the baseline reading) will be managed by administration of ephedrine 15 mg Reactive hypertension (defined as systolic blood pressure ≥120% from the baseline reading) will be managed (if persisted > 1-reading) by stoppage of the infusion till the next systolic blood pressure reading.

Intraoperative bradycardia (defined as heart rate less than 55 bpm) will be managed by stoppage of the vasopressor infusion if not associated with hypotension. The infusion will be then re-started in a reduced rate (50%) when the heart rate is more than 55 bpm. IV atropine bolus (0.5 mg) will be administered if bradycardia persisted despite stoppage of the infusion. If accompanied with hypotension, bradycardia will be managed by IV bolus of ephedrine 9 mg.

Reactive tachycardia (heart rate >130% of baseline) not related to hypotension or ephedrine infusion, will be managed if persisted by stoppage of the infusion. The infusion will be then re-started in a reduced rate (50% of the initial dose) when heart rate will have decreased to be within 30% of the baseline reading.

Fluid administration will be continued up to a maximum of 1.5 liters. After delivery, an oxytocin bolus (0.5 IU) will be delivered over five seconds, followed by infusion at a rate of 2.5 IU/hour.

ELIGIBILITY:
Inclusion Criteria:

* full-term singleton pregnant women, admitted for elective cesarean delivery

Exclusion Criteria:

* Patients with uncontrolled cardiac morbidities (patients with tight valvular lesion, impaired contractility with ejection fraction < 50%, heart block, and arrhythmias),
* hypertensive disorders of pregnancy,
* peripartum bleeding,
* coagulation disorders (patients with INR >1.4 and or platelet count < 80000 /dL) or any contraindication to regional anesthesia,
* baseline systolic blood pressure (SBP) < 100 mmHg

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 212 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
incidence of post-spinal hemodynamic instability | 1 min after spinal anesthesia until 5 min after the delivery
  the occurrence of either, hypotension, hypertension, bradycardia, and/or tachycardia

SECONDARY OUTCOMES:
umbilical pH | 5 min after delivery
  from umbilical artery
Apgar | 5 min after delivery
  assessment of Breathing effort, Heart rate, Muscle tone, Reflexes, Skin color; Each category is scored with 0, 1, or 2
heart rate | 1 min after spinal anesthesia until 5 min after the delivery
  beat/min
systolic blood pressure | 1 min after spinal anesthesia until 5 min after the delivery
  mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are available from the authors upon reasonable request.